CLINICAL TRIAL: NCT04179409
Title: A 48-Week, Open Label, Study to Evaluate the Efficacy and Safety of AMONDYS 45, EXONDYS 51, VYONDYS 53 in Subjects With DuchenneMuscular Dystrophy Carrying Eligible DMD Duplications.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kevin Flanigan (Other)
Collaborators: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Kevin Flanigan, Professor of Neurology, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRPT-Dup-US-001
Record Dates: First submitted 2019-08-12; First posted 2019-11-27 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD; Exon Skipping
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — casimersen; eteplirsen; golodirsen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AMONDYS 45 (Experimental): This arm will involve the treatment of boys with DMD who have a duplication of exon 45, for which AMONDYS 45 will target skipping of this exon.
  Interventions: Drug: Amondys 45
- EXONDYS 51 (Experimental): This arm will involve the treatment of boys with DMD who have a duplication of exon 51, for which EXONDYS 51 will target skipping of this exon.
  Interventions: Drug: Exondys 51
- VYONDYS 53 (Experimental): This arm will involve the treatment of boys with DMD who have a duplication of exon 53, for which VYONDYS 53 will target skipping of this exon.
  Interventions: Drug: Vyondys 53

INTERVENTIONS:
Drug: Amondys 45 — This drug is used to target skipping of exon 45 of the dystrophin gene.
  Other Names: SRP-4045; Casimersen
  Arms: AMONDYS 45
Drug: Exondys 51 — This drug is used to target skipping of exon 51 of the dystrophin gene.
  Other Names: Eteplirsen; AVI-4658
  Arms: EXONDYS 51
Drug: Vyondys 53 — This drug is used to target skipping of exon 53 of the dystrophin gene.
  Other Names: SRP-4053; Golodirsen
  Arms: VYONDYS 53

SUMMARY:
This is an 48-week open-label study to determine the efficacy and safety of AMONDYS 45, EXONDYS 51, VYONDYS 53 for the treatment of boys with duchenne muscular dystrophy who have a single exon duplication of either exon 45, 51 or 53, respectively. There will be weekly infusions and two muscle biopsies at baseline and at month 12.

DETAILED DESCRIPTION:
DMD is a rare, serious, debilitating, and ultimately fatal, disease for which there is an urgent need to develop safe and effective therapies. In order to efficiently meet this urgency and the needs of the subject community, the study evaluates the efficacy and safety of AMONDYS 45, EXONDYS 51, VYONDYS 53 administration over approximately 1 year in DMD subjects with duplication mutations amenable to treatment by exon 45, 51 or exon 53 skipping. Skipping of a single copy of the duplicated exon is expected to result in a wild-type (WT) DMD transcript allowing the expression of a WT, full length dystrophin protein. Successful skipping of a single copy of the duplicated exon in in vitro and in vivo models has been reported in the literature. AMONDYS 45, EXONDYS 51, VYONDYS 53 have the potential to be disease-modifying treatments for boys with DMD mutations amenable to exon 45, 51 and exon 53 skipping, respectively.

The totality of the non-clinical data with these PMOs as well as AVI-4225 (targeting exon 23) and EXONDYS 51 suggests that PMOs are well tolerated in the non-clinical setting. Moreover, treatment with EXONDYS 51(at 30 mg/kg and 50 mg/kg) has been well-tolerated by boys with DMD deletion mutations amenable to skipping exon 51. The relatively low expected risk for subjects exposed to AMONDYS 45, EXONDYS 51, VYONDYS 53 and the urgent medical need for a treatment for this subject population support the conclusion that the potential benefits of exposing subjects to AMONDYS 45, EXONDYS 51, VYONDYS 53 outweigh the potential risks.

ELIGIBILITY:
Inclusion Criteria:

* Is a male with DMD and has an out-of-frame duplication of either exon 45, 51, or 53, with a normal copy number of all other DMD exons.
* Is above age 6 months of age.
* Has sufficient muscle mass in a pair of bilateral muscles that will allow for pre- and post-treatment muscle biopsies per PI discretion.
* If the subject is ambulant and 4 years old or greater and has been on a stable dose or dose equivalent of oral corticosteroids for at least 12 weeks prior to Week 1 the dose is expected to remain constant (except for modifications to accommodate changes in weight) throughout the study.

Exclusion Criteria:

* Any additional missing exon for DMD that cannot be treated with study drugs.

Other inclusion/exclusion criteria apply

Min Age: 6 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Flanigan, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Aartsma-Rus A, Fokkema I, Verschuuren J, Ginjaar I, van Deutekom J, van Ommen GJ, den Dunnen JT. Theoretic applicability of antisense-mediated exon skipping for Duchenne muscular dystrophy mutations. Hum Mutat. 2009 Mar;30(3):293-9. doi: 10.1002/humu.20918. PMID 19156838
- [Background] Greer KL, Lochmuller H, Flanigan K, Fletcher S, Wilton SD. Targeted exon skipping to correct exon duplications in the dystrophin gene. Mol Ther Nucleic Acids. 2014 Mar 18;3(3):e155. doi: 10.1038/mtna.2014.8. PMID 24643206
- [Background] Mendell JR, Rodino-Klapac LR, Sahenk Z, Roush K, Bird L, Lowes LP, Alfano L, Gomez AM, Lewis S, Kota J, Malik V, Shontz K, Walker CM, Flanigan KM, Corridore M, Kean JR, Allen HD, Shilling C, Melia KR, Sazani P, Saoud JB, Kaye EM; Eteplirsen Study Group. Eteplirsen for the treatment of Duchenne muscular dystrophy. Ann Neurol. 2013 Nov;74(5):637-47. doi: 10.1002/ana.23982. Epub 2013 Sep 10. PMID 23907995
- [Background] Mendell JR, Goemans N, Lowes LP, Alfano LN, Berry K, Shao J, Kaye EM, Mercuri E; Eteplirsen Study Group and Telethon Foundation DMD Italian Network. Longitudinal effect of eteplirsen versus historical control on ambulation in Duchenne muscular dystrophy. Ann Neurol. 2016 Feb;79(2):257-71. doi: 10.1002/ana.24555. Epub 2016 Jan 8. PMID 26573217

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AMONDYS 45 | EXONDYS 51 | VYONDYS 53
Started | 2 | 0 | 1
Completed | 2 | 0 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: We did not enroll any participants in the EXONDYS 51 treatment arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | AMONDYS 45 | EXONDYS 51 | VYONDYS 53 | Total
Number analyzed (Participants) | 2 | 0 | 1 | 3
Age, Customized [Mean (Standard Deviation); unit: Years]
  Age | 12 (6) |  | 23 (0) | 16 (7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 2 |  | 1 | 3
  Female | 0 |  | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  | 0 | 1
  Not Hispanic or Latino | 1 |  | 1 | 2
  Unknown or Not Reported | 0 |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 | 0
  Asian | 0 |  | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0
  Black or African American | 0 |  | 0 | 0
  White | 2 |  | 1 | 3
  More than one race | 0 |  | 0 | 0
  Unknown or Not Reported | 0 |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Dystrophin Expression From Baseline Following Treatment With Either AMONDYS 45 (Previously Casimersen), EXONDYS 51 (Previously Eteplirsen ), or VYONDYS 53 (Previously Golodirsen)
Description: This will be assessed by the comparison of quantification of protein in muscle biopsy tissue by western blot from baseline to 1 year post-initiation of treatment.
Time Frame: Baseline, 1 year
Population: We did not enroll any participants in the EXONDYS 51 treatment arm.
Measure: Mean (Standard Deviation); unit: Percent of Healthy Control
Arm/Group | AMONDYS 45 | EXONDYS 51 | VYONDYS 53
Number analyzed (Participants) | 2 | 0 | 1
Percent of Healthy Control | 3.1 (1.8) |  | 6.1 (0)

2. Primary Outcome: Monitoring for the Development of Unacceptable Toxicity.
Description: This will be measured by capturing and reviewing Adverse Events as defined by CTCAE v4.0.
Time Frame: 1 year
Population: We did not enroll any participants in the EXONDYS 51 treatment arm.
Measure: Number; unit: Events
Arm/Group | AMONDYS 45 | EXONDYS 51 | VYONDYS 53
Number analyzed (Participants) | 2 | 0 | 1
Events | 17 |  | 11

3. Secondary Outcome: Change in Dystrophin Expression From Baseline Following Treatment With Either AMONDYS 45 (Previously Casimersen), EXONDYS 51 (Previously Eteplirsen ), or VYONDYS 53 (Previously Golodirsen).
Description: This will be assessed by the comparison of immunofluorescent staining in muscle biopsy tissue from baseline to 1 year post-initiation of treatment.
Time Frame: 1 year
Population: We did not enroll any participants in the EXONDYS 51 treatment arm.
Measure: Mean (Standard Deviation); unit: % Dystrophin Postive Fibers
Arm/Group | AMONDYS 45 | EXONDYS 51 | VYONDYS 53
Number analyzed (Participants) | 2 | 0 | 1
% Dystrophin Postive Fibers | 38 (25) |  | 30.8 (0)

ADVERSE EVENTS:
Time Frame: Data was collected over 1 year.
Description: We did not enroll any participants in the EXONDYS 51 treatment arm.
Arm/Group | AMONDYS 45 | EXONDYS 51 | VYONDYS 53
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 0/0 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMONDYS 45 (N=2) | EXONDYS 51 (N=0) | VYONDYS 53 (N=1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Procedural Discomfort (General disorders) | 2 (4) | 0 (0) | 1 (3)
Kidney Stones (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Bruising (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Procedural Discomfort (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Wound Dihiscence (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Laceration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Correction of a Congenital Defect (General disorders) | 1 (1) | NA | 0 (0)
Non-Procedural Discomfort (General disorders) | 1 (3) | NA | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT04179409/Prot_SAP_000.pdf